CLINICAL TRIAL: NCT02537782
Title: Investigating Inhomogeneities of Regional Myocardial WORKload and Metabolism in a Cardiac Resynchronisation Therapy Patient Population
Brief Title: Myocardial Work and Metabolism in CRT
Acronym: WORK-CRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, prof. dr. Jens-Uwe Voigt, prof. dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S538235_v1.2
Record Dates: First submitted 2015-08-12; First posted 2015-09-02 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Left Ventricular Dyssynchrony; Heart Failure; Left Bundle Branch Block; Cardiomyopathy
Keywords: Cardiac Resynchronisation Therapy; Heart Failure; Left ventricular dyssynchrony; Echocardiography; Apical rocking; Septal flash
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block; Cardiomyopathies | interventions — Cardiac Resynchronization Therapy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiac resynchronisation therapy implantation (Other): Patients with current guideline-based indication for CRT implantation.
  Interventions: Device: Cardiac resynchronisation therapy; Other: Echocardiography; Other: Magnetic Resonance Imaging; Other: Positron Emission Tomography

INTERVENTIONS:
Device: Cardiac resynchronisation therapy
Other: Echocardiography
Other: Magnetic Resonance Imaging
Other: Positron Emission Tomography

SUMMARY:
Several attempts have been made to refine selection criteria for cardiac resynchronisation therapy (CRT) in heart failure patients with reduced ejection fraction (HFrEF). Previously proposed parameters probably do not sufficiently reflect the underlying mechanical dyssynchrony of the left ventricle (LV). Earlier work of our research group suggests that better candidate selection can rely on the direct observation or measurement of this LV mechanical dyssynchrony by means of non-invasive imaging. In this study apical rocking and other non-invasive measures of LV mechanical dyssynchrony will be applied to evaluate regional myocardial workload and metabolism, and determine their predictive value in CRT response.

ELIGIBILITY:
Inclusion Criteria

Subject is eligible for CRT implantation according to current European Society of Cardiology guidelines of 2013.

* The patient should receive guideline-directed optimal medical therapy for heart failure and left ventricular (LV) function must be severely depressed (LV ejection fraction ≤35%).
* The patients should be in NYHA functional class II, III or ambulatory IV.
* The patient should present a left bundle branch block (LBBB) with QRS duration of >120ms or a non-LBBB with QRS >150ms.
* Also patients with conventional pacemaker in NYHA functional class III and ambulatory IV if high percentage of ventricular pacing, are eligible for CRT implantation.
* Subject is in stable sinus rhythm at the time of CRT implant and during the last 2 weeks prior to inclusion.
* Subject is 18 years or older and able and willing to consent.

Exclusion Criteria:

* Impossible to obtain LV volumes by echocardiography.
* Right bundle branch block.
* Permanent atrial fibrillation, flutter or tachycardia (>100 bpm).
* Recent myocardial infarction, within 40 days prior to enrolment.
* Subject underwent coronary artery bypass graft (CABG) or valve surgery, within 90 days.
* Post heart transplantation, or is actively listed on the transplantation list, or has reasonable probability (per investigator's discretion) of undergoing transplantation in the next year.
* Implanted with a LV assist device (LVAD), or has reasonable probability (per investigator's discretion) of receiving a LVAD in the next year.
* Severe aortic stenosis (with a valve area of <1.0 cm2 or significant valve disease expected to be operated on within study period).
* Complex and uncorrected congenital heart disease.
* Breastfeeding women, women of child bearing potential.
* Enrolled in one or more concurrent studies that would confound the results of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-12-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac resynchronisation therapy (CRT) response assessed by echocardiography | Change of left ventricular end-systolic volume (LVESV) between baseline and 6 months after CRT implantation
  Reduction in LVESV ≥15% from baseline
CRT response assessed by echocardiography | Change of LVESV between baseline and 12 months after CRT implantation
  Reduction in LVESV ≥15% from baseline

SECONDARY OUTCOMES:
Reverse left ventricular remodelling measured as changes in left ventricular volume by echocardiography | Change of remodelling between baseline, 6 and 12 months after CRT implantation
  Measured as changes in left ventricular volume by echocardiography
Reverse left ventricular remodelling measured as changes in left ventricular ejection fraction by echocardiography | Change of remodelling between baseline, 6 and 12 months after CRT implantation
  Measured as changes in left ventricular ejection fraction by echocardiography
New York Heart Association (NYHA) class changes | Change of NYHA class between baseline, 6 and 12 months after CRT implantation
  A decrease of ≥1 NYHA class
Functional capacity changes assessed by 6-minute walking test | Change of functional capacity between baseline and 6 months after CRT implantation
  Assessed by 6-minute walking test
Functional capacity changes assessed by peak oxygen uptake ergospirometry (VO2max) | Change of functional capacity between baseline and 6 months after CRT implantation
  Assessed by peak oxygen uptake ergospirometry (VO2max)
Quality of Life changes | Change of QoL between baseline, 6 and 12 months after CRT implantation
Heart failure related hospital admissions | Assessment of the number of hospital admissions at 6 and 12 months after CRT implantation
Death | Assessment of possible death at 6 and 12 months after CRT implantation
  Death by heart failure, sudden cardiac death and all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Uwe Voigt, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Otto A Smiseth, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Degtiarova G, Claus P, Duchenne J, Cvijic M, Schramm G, Nuyts J, Voigt JU, Gheysens O. Low septal to lateral wall 18F-FDG ratio is highly associated with mechanical dyssynchrony in non-ischemic CRT candidates. EJNMMI Res. 2019 Dec 9;9(1):105. doi: 10.1186/s13550-019-0575-9. PMID 31820130